CLINICAL TRIAL: NCT04294498
Title: A Phase II Study of Durvalumab (MEDI 4736) for Advanced Hepatocellular Carcinoma in Patients With Active Chronic Hepatitis B Virus Infection
Brief Title: Durvalumab for Advanced Hepatocellular Carcinoma in Patients With Active Chronic Hepatitis B Virus Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201910075MIPD
Record Dates: First submitted 2020-02-25; First posted 2020-03-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Checkpoint inhibitor; Hepatocellular carcinoma; Chronic Hepatitis B
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B, Chronic | interventions — durvalumab; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durvalumab (Experimental): Durvalumab
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Entecavir treatment for chronic hepatitis B will be started within one week before initiation of durvalumab treatment for advanced hepatocellulcar carcinoma
  Other Names: Entecavir

SUMMARY:
PD1 blockade has been approved as salvage therapy for advanced hepatocellular carcinoma (HCC). Although there is not solid evidence that PD1 blockade would induce hepatitis B virus (HBV) reactivation, previous clinical trials of PD1 blockade required enrolled patients to receive anti-HBV medications and control the viral load to be under 100-2000 IU/mL before initiation of PD1 blockade therapy. Such a requirement may not be necessary and could delay the treatment. Guidelines for prevention of chemotherapy induced HBV reactivation only suggest combining anti-HBV medications during the chemotherapy course without such a requirement of very load HBV viral load.

The investigators hypothesized that under anti-HBV medications, patients with advanced HCC and active chronic hepatitis B virus (HBV) infection can receive durvalumab treatment without increased risks of HBV reactivation and related complications.

DETAILED DESCRIPTION:
Although durvalumab has not been approved as treatment for HCC, similar PD1 blockade agents such as nivolumab and pembrolizumab have gain approval as salvage therapy for advanced HCC. The investigators will enroll 43 patients with active (defined as serum viral load > 2000 IU/mL) chronic HBV infection (defined as positive serum HBV surface antigen). All patients would receive entecavir within 7 days of initiation of durvalumab treatment. Durvalumab 1500 mg would be given intravenously every 4 weeks until confirmed disease progression, intolerable side effects, or completion of 24 treatment. Tumor assessment will be performed every 8-12 weeks. HBV viral load will be monitored at least once per month. Entecavir treatment will be continued at least 6 months after discontinuation of durvalumab treatment.

ELIGIBILITY:
Inclusion criteria

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Histologically or clinically (typical HCC imaging findings by multi-phase CT or MRI) diagnosed HCC.
* Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy.
* HBeAg (-) active chronic HBV infection, defined by positive serum HBsAg AND serum HBV DNA ≥ 2,000 IU/mL.
* No previous immune checkpoint inhibitor treatment
* The patient refuses, has disease progression on, or does not tolerate treatment kinase inhibitors such as sorafenib or lenvatinib
* Age > 20 years at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Child-Pugh class A
* ≥1 measurable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Body weight >30 kg
* Adequate normal organ and marrow function as defined below:

  1. Haemoglobin ≥9.0 g/dL
  2. Absolute neutrophil count (ANC) ≥1.0 x 109/L (> 1,000 per mm3)
  3. Platelet count ≥75 x 109/L (>75,000 per mm3)
  4. Serum bilirubin ≤2 x institutional upper limit of normal (ULN).
  5. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless active liver malignancies are present, in which case it must be ≤5x ULN
  6. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks

Exclusion criteria

* Serum HBeAg (+)
* Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
* Active or prior documented GI variceal bleed or history of upper GI bleeding, ulcers, or esophageal varices with bleeding within 12 months; adequate endoscopic therapy according to institutional standards is required for patients with history of esophageal variceal bleeding or assessed as high risk for esophageal variceal by the treating investigator.
* Previous organ transplants
* Participation in another clinical study with an investigational product during the last 2 weeks
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤14 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by the principal investigator
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection (except HBV infection), symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
* History of active primary immunodeficiency or HIV infection
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), and hepatitis C
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The rate of HBV reactivation during durvalumab treatment | 30 months
  To assess the rate of HBV reactivation during durvalumab treatment, defined as a ≥2 log (100-fold) increase in serum HBV DNA compared to the baseline level.

SECONDARY OUTCOMES:
The rate of hepatitis flare during durvalumab treatment | 30 months
  To assess the rate of hepatitis flare, defined as an ALT increase to ≥3 times the baseline level and >100 U/L, during durvalumab treatment.
To assess the rate of HBV-associated hepatitis during durvalumab treatment. | 30 months
  To assess the rate of HBV-associated hepatitis, defined as HBV reactivation plus hepatitis flare, during durvalumab treatment.
To assess the efficacy of durvalumab treatment | 30 months
  To assess the efficacy of durvalumab treatment, as determined by the objective tumor response rates per RECIST v1.1.
To assess the efficacy of durvalumab treatment | 30 months
  To assess the efficacy of durvalumab treatment, as determined by time to tumor progression.
To assess the efficacy of durvalumab treatment | 30 months
  To assess the efficacy of durvalumab treatment, as determined by progression-free survival.
To assess the efficacy of durvalumab treatment | 30 months
  To assess the efficacy of durvalumab treatment, as determined by overall survival.
To assess the adverse events during durvalumab treatment. | 30 months
  To assess the adverse events, defined by CTC-AE version 5.0, during durvalumab treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Shao YY, Chen CT, Chuang CH, Su TH, Ho MC, Tseng TC, Liu TH, Wu TC, Cheng AL, Hsu CH. Prompt initiation of durvalumab and tremelimumab for unresectable hepatocellular carcinoma in patients with chronic active hepatitis B: a phase 2 clinical trial. Br J Cancer. 2025 May;132(9):822-827. doi: 10.1038/s41416-025-02978-7. Epub 2025 Mar 24. PMID 40128285